CLINICAL TRIAL: NCT03056794
Title: Natural History and Advanced Genetic Study of Pyruvate Dehydrogenase Complex Deficiencies (North American Mitochondrial Disease Consortium, Rare Diseases Clinical Research Network, Project 7413)
Brief Title: Natural History and Advanced Genetic Study of Pyruvate Dehydrogenase Complex Deficiencies
Status: Recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Rare Diseases Clinical Research Network (Network); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Jirair Krikor Bedoyan, Associate Professor, University of Pittsburgh
Other Study IDs: STUDY21090146; 5U54NS078059-05 (NIH)
Record Dates: First submitted 2017-01-27; First posted 2017-02-17 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Pyruvate Dehydrogenase Complex Deficiency Disease
Keywords: pyruvate; pyruvate dehydrogenase; PDC; PDCD
MeSH Terms: conditions — Pyruvate Dehydrogenase Complex Deficiency Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood sample for DNA and biochemical analysis. Saliva, buccal swab, urine sample, blood sample, or skin sample for NAMDC biorepository (optional).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PDC Deficiency: Pyruvate Dehydrogenase Complex Deficiency Disease
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study. The investigators will collect data about exposure to responses to dietary supplements, medications, and the ketogenic diet.

SUMMARY:
Children and adults with pyruvate dehydrogenase complex deficiency (PDCD) are participating in a research study seeking to better understand the genetic causes, symptoms, usefulness of current treatments, and outcomes for these disorders. The research project involves completing a questionnaire about the individual or family's medical history and experiences with PDCD, review of medical records by the researchers, and in some cases, advanced genetic testing.

DETAILED DESCRIPTION:
Pyruvate dehydrogenase complex deficiencies (PDCDs) are a major class of mitochondrial diseases, limiting oxidation of carbohydrate for energy production, which is especially important in the brain. So far, there is not a definitive treatment for these disorders. This study, "Advanced Genetic Study and Pilot Newborn Screening for Disorders of Pyruvate Metabolism," will continue with the created database with information that is collected over a long period of time about patients with PDCDs. This database is part of the existing North American Mitochondrial Disease Consortium (NAMDC) Patient Data Registry and Biorepository database. The study will collect data specific to PDC deficiencies, including data that is derived from patients/families. Approximately 75 subjects with confirmed PDCD will be enrolled over 5 years. The genetic basis and pathophysiology will be explored in up to a third of confirmed PDC deficient patients, who currently have not been found to have an identified mutation in DLD or any of the five "primary" PDC-specific genes (PDHA1, PDHB, DLAT, PDHX, and PDP1), and who might benefit from different treatments.

The specific aims of the study are:

1. Continue to add to the Pyruvate Dehydrogenase Complex Deficiencies (PDCDs) specific database within the NAMDC Patient Data Registry
2. Use advanced genetic analysis technologies to find mutations in those people in whom none has been found

About this Study:

This study will collect comprehensive longitudinal natural history clinical data for proven Pyruvate Dehydrogenase Complex deficiencies (PDCDs), including data about diagnoses, symptoms, and outcomes. The study will include data from patients/parents as well as medical data. The investigators will use medical records and a short questionnaire targeted to collect information about critical outcomes. This questionnaire will collect information from the subject and parent about the importance of different outcomes and allow families to discuss other outcomes that they may consider important at home. Additional details of treatment will be sought to maximize our knowledge about their effects and serve to inform future clinical trials.

Data Dictionary: On file at Data Monitoring Core Council in Cincinnati Children's Hospital Medical Center and has been provided to investigators at University Hospitals Cleveland Medical Center.

ELIGIBILITY:
Inclusion Criteria:

1. Low PDC activity in skin fibroblasts, blood lymphocytes or a muscle biopsy, below the reference range, and with valid internal controls to establish sample and assay integrity, and have had PDHA1 testing, and/or
2. A known pathogenic mutation of a gene associated with PDC deficiency.

Relative Subjects Inclusion Criteria:

1. First or second degree relative of a primary subject for whom genetic testing indicates the presence of variants of unknown significance (VUS).

Exclusion Criteria:

1. Another chronic neurological disease (mitochondrial or non-mitochondrial) which is not considered likely to be related to PDC deficiency.
2. Inadequacy of needed blood or tissue sample and unwillingness or inability to submit such a sample.
3. Unwillingness to participate in the NAMDC Patient Data Registry and Biorepository protocol.

Relative Subjects Exclusion Criteria:

1. Inadequacy of needed blood sample and unwillingness or inability to submit such a sample.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children and adults with pyruvate dehydrogenase complex deficiency
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Survival outcomes in pyruvate dehydrogenase deficiency disease | Data will be collected about duration of survival from birth until the last date known to be living at the time of data analysis.
  Survival will be measured in years and months.

SECONDARY OUTCOMES:
Neurological outcomes in pyruvate dehydrogenase deficiency disease | Through a participant questionnaire and retrospective review of medical records, neurological outcomes will be assessed for the entire lifetime of the participant up to the time of data collection.
  The number of participants with each neurological outcome will be assessed by analyzing questionnaire and medical record data. Neurological outcomes include, but are not limited to, developmental delay/intellectual disability, seizures, muscle weakness and abnormalities of tone, ataxia, neuropathy, dysautonomia, involuntary movements, microcephaly, hearing loss, and ophthalmologic abnormalities/ vision impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Jirair K. Bedoyan, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data to be submitted to dbGap, as well as NAMDC researchers and the RDCRN.

REFERENCES:
- [Background] DeBrosse SD, Okajima K, Zhang S, Nakouzi G, Schmotzer CL, Lusk-Kopp M, Frohnapfel MB, Grahame G, Kerr DS. Spectrum of neurological and survival outcomes in pyruvate dehydrogenase complex (PDC) deficiency: lack of correlation with genotype. Mol Genet Metab. 2012 Nov;107(3):394-402. doi: 10.1016/j.ymgme.2012.09.001. Epub 2012 Sep 7. PMID 23021068
- [Background] Huang X, Bedoyan JK, Demirbas D, Harris DJ, Miron A, Edelheit S, Grahame G, DeBrosse SD, Wong LJ, Hoppel CL, Kerr DS, Anselm I, Berry GT. Succinyl-CoA synthetase (SUCLA2) deficiency in two siblings with impaired activity of other mitochondrial oxidative enzymes in skeletal muscle without mitochondrial DNA depletion. Mol Genet Metab. 2017 Mar;120(3):213-222. doi: 10.1016/j.ymgme.2016.11.005. Epub 2016 Nov 12. PMID 27913098
- [Background] Bedoyan JK, Yang SP, Ferdinandusse S, Jack RM, Miron A, Grahame G, DeBrosse SD, Hoppel CL, Kerr DS, Wanders RJA. Lethal neonatal case and review of primary short-chain enoyl-CoA hydratase (SCEH) deficiency associated with secondary lymphocyte pyruvate dehydrogenase complex (PDC) deficiency. Mol Genet Metab. 2017 Apr;120(4):342-349. doi: 10.1016/j.ymgme.2017.02.002. Epub 2017 Feb 2. PMID 28202214
- [Background] Ferdinandusse S, Friederich MW, Burlina A, Ruiter JP, Coughlin CR 2nd, Dishop MK, Gallagher RC, Bedoyan JK, Vaz FM, Waterham HR, Gowan K, Chatfield K, Bloom K, Bennett MJ, Elpeleg O, Van Hove JL, Wanders RJ. Clinical and biochemical characterization of four patients with mutations in ECHS1. Orphanet J Rare Dis. 2015 Jun 18;10:79. doi: 10.1186/s13023-015-0290-1. PMID 26081110
- [Background] Deeb KK, Bedoyan JK, Wang R, Sremba L, Schroeder MC, Grahame GJ, Boyer M, McCandless SE, Kerr DS, Zhang S. Somatic mosaicism for a novel PDHA1 mutation in a male with severe pyruvate dehydrogenase complex deficiency. Mol Genet Metab Rep. 2014 Aug 28;1:362-367. doi: 10.1016/j.ymgmr.2014.08.001. eCollection 2014. PMID 27896109
- [Background] Shin HK, Grahame G, McCandless SE, Kerr DS, Bedoyan JK. Enzymatic testing sensitivity, variability and practical diagnostic algorithm for pyruvate dehydrogenase complex (PDC) deficiency. Mol Genet Metab. 2017 Nov;122(3):61-66. doi: 10.1016/j.ymgme.2017.09.001. Epub 2017 Sep 8. PMID 28918066
- [Background] Bedoyan JK, Hecht L, Zhang S, Tarrant S, Bergin A, Demirbas D, Yang E, Shin HK, Grahame GJ, DeBrosse SD, Hoppel CL, Kerr DS, Berry GT. A novel null mutation in the pyruvate dehydrogenase phosphatase catalytic subunit gene (PDP1) causing pyruvate dehydrogenase complex deficiency. JIMD Rep. 2019 Jun 17;48(1):26-35. doi: 10.1002/jmd2.12054. eCollection 2019 Jul. PMID 31392110